CLINICAL TRIAL: NCT04945655
Title: Impact of a School- and Primary Care-based Multicomponent Intervention on HPV Vaccination Acceptability Among French Adolescents: a Cluster Randomized Controlled Trial
Brief Title: Impact of a School- and Primary Care-based Multicomponent Intervention on HPV Vaccination Acceptability
Acronym: PrevHPV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: C20-76; 2020-A02031-38 (Registry Identifier: ID-RCB)
Record Dates: First submitted 2021-06-07; First posted 2021-06-30 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2023-07

CONDITIONS: HPV Vaccine Acceptability
Keywords: Human Papillomavirus; Vaccination coverage; eHealth tools; Motivational interview; Pragmatic randomized controlled trial; Effectiveness; Implementation; Vaccination behaviors

STUDY DESIGN:
Intervention Model Description: Multicentre cluster randomized controlled trial using an incomplete factorial design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Arm 1: component 1 + component 2 + component 3 (Experimental): Adolescents and parents' education and motivation at school (component 1) + General practitioners' training (component 2) + Access to vaccination at school (component 3)
  Interventions: Other: Adolescents and parents' education and motivation at school (component 1); Other: General practitioners' training (component 2); Other: Access to vaccination at school (component 3)
- Arm 2: component 1 + component 2 (Experimental): Adolescents and parents' education and motivation at school (component 1) + General practitioners' training (component 2)
  Interventions: Other: Adolescents and parents' education and motivation at school (component 1); Other: General practitioners' training (component 2)
- Arm 3: component 1 + component 3 (Experimental): Adolescents and parents' education and motivation at school (component 1) + Access to vaccination at school (component 3)
  Interventions: Other: Adolescents and parents' education and motivation at school (component 1); Other: Access to vaccination at school (component 3)
- Arm 4: component 1 (Experimental): Adolescents and parents' education and motivation at school (component 1)
  Interventions: Other: Adolescents and parents' education and motivation at school (component 1)
- Arm 5: component 2 (Experimental): General practitioners' training (component 2)
  Interventions: Other: General practitioners' training (component 2)
- Arm 6: Control (No Intervention): No intervention

INTERVENTIONS:
Other: Adolescents and parents' education and motivation at school (component 1) — The component 1 includes first an information group session (duration: 1h30) on HPV infection and vaccination for parents. This session starts with a webconference delivered by two medical experts on HPV, using a standardized presentation. Then, a discussion is open for parents' questions and/or comments.
  Second, adolescents participate during the school time to two educational group sessions on HPV infections and vaccination, using a pedagogy based on active learning. These sessions (duration: 2h each) are delivered by the school staff (e.g., nurse, teacher in life sciences) using an educational package comprising: a guide that describes activities that should be implemented during each session; one video and a fact sheet developed by health students; a serious video game that promotes HPV vaccination and accessible on an internet website. Before the sessions, the school staff is encouraged to attend an e-learning training course (duration: 1 hour).
  Arms: Arm 1: component 1 + component 2 + component 3; Arm 2: component 1 + component 2; Arm 3: component 1 + component 3; Arm 4: component 1
Other: General practitioners' training (component 2) — The component 2 consists of an individual e-learning training session for general practitioners (GPs) that is accessible on computer and smartphone. Lasting 3 hours, GPs are able to access to the training whenever they want and then to progress at their own pace. The training includes three main parts: up-dated information on HPV infection and vaccination; an introduction to the use of motivational interviewing techniques in the field of vaccination; and a presentation of the decision aid tool developed as part of the intervention and explanation of how to use it during consultations. GPs may ask questions to the consortium team by using a dedicated chat.
  Arms: Arm 1: component 1 + component 2 + component 3; Arm 2: component 1 + component 2; Arm 5: component 2
Other: Access to vaccination at school (component 3) — The component 3 aims at enhancing access to HPV vaccination for adolescents by offering them the first free-of-charge injection at school, without any medical prescription. For each concerned school, we organise a vaccination day inside the school premises where health professionals (one physician and one nurse) from the local vaccination centre initiate HPV vaccination with Gardasil-9® (in accordance with the French recommendations) for all eligible adolescents.
  Arms: Arm 1: component 1 + component 2 + component 3; Arm 3: component 1 + component 3

SUMMARY:
This study aims at evaluating the effectiveness, efficiency and implementation of a multicomponent intervention (components being applied in combination or alone) on the acceptability of HPV vaccine among French adolescents (11-14 years old) through a cluster randomized controlled trial. The primary outcome to measure acceptability is vaccine coverage. The three components are: adolescents and parents' education and motivation at school (component 1); general practitioners' training (component 2); and access to vaccination at school (component 3). Ninety municipalities are included and randomized into six groups of 15 municipalities, according an incomplete factorial plan.

ELIGIBILITY:
Adolescents and parents' education and motivation at school (component 1 -- arms 1-4) and "KABP-6C" survey among adolescents and parents (arms 1-6)

Inclusion Criteria:

* Adolescents (school years 9-10), and parents of adolescents (school years 7-10) attending secondary schools in the participating municipalities.

Exclusion Criteria:

* /

General practitioners' training (component 2) and "KABP-6C" survey among general practitioners (arms 1, 2 and 5)

Inclusion Criteria:

* General practitioners' practicing in the participating municipalities.

Exclusion Criteria:

* Exclusive particular type of practice.
* Planning to retire or move their practice within the study period.
* No internet access.

Access to vaccination at school (component 3 -- arms 1 and 3)

Inclusion Criteria:

* Adolescents (school years 7-10) attending secondary schools in the participating municipalities, aged 11-14 years (with a possible catch-up for those aged 15-19 years according to the French recommendations).

Exclusion Criteria:

* Having initiated HPV vaccination.
* No written consent from parents/caregivers for vaccination.
* Contraindication to HPV vaccination.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 30739 (Actual)
Dates: Start 2021-11-15 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2023-04-30 (Actual)

PRIMARY OUTCOMES:
HPV vaccine coverage (≥ 1 dose) | 2 months after intervention
  Percentage of adolescents aged 11-14 years, living in the municipality, who have received at least one dose of HPV vaccine

SECONDARY OUTCOMES:
HPV vaccine coverage (≥ 1 dose) | 6 months and 12 months after intervention
  Percentage of adolescents aged 11-14 years, living in the municipality, who have received at least one dose of HPV vaccine
HPV vaccine coverage (2 doses) | 2 months, 6 months and 12 months after intervention
  Percentage of adolescents aged 11-14 years, living in the municipality, who have received two doses of HPV vaccine
HPV vaccination intention | Before intervention and 2 months after intervention
  Percentage of each group of participants (adolescents, parents and general practitioners) who have the intention to initiate/have their child vaccinated/recommend HPV vaccination
Knowledge, attitude, beliefs and practices towards HPV vaccination and psychological determinants of vaccination intention ("KABP-6C") | Before intervention and 2 months after intervention
  Each group participants' (adolescents, parents and general practitioners) knowledge and attitude towards HPV vaccination will be assessed for each of the " 6-C " components (Confidence, Complacency, Constraints, Calculation, Collective responsibility and social Conformism). Following results from otherwise onging research on psychological antecedents of vaccination, a 7 th C has been identified, refering to Confidence in the system (including reactance). The 6C thus has been extended to a 7C scale.
  In addition to analysis of individual items, a score of knowledge (from 0 - poor knowledge -- to 12 -- good knowledge) and a score of attitude (from 0 - unfavourable attitude -- to 24 - very favourable attitude) will then be calculated. Practices towards HPV vaccination (self-declared vaccination status / recommendation to patients) will be assessed using closed questions. Data will be collected using ad hoc self-administered online KABP-7C questionnaires.
Incremental Cost-Effectiveness Ratio | 2 months after intervention
  Incremental Cost-Effectiveness Ratio
Intervention components' dose and fidelity | Intervention components' implementation period
  Number of different activities really performed for each component / number of activities planned for each component according to the protocol. Data come from regular activity reports collected on a standardised form during components' implementation.
Reached populations | Intervention components' implementation period
  Percentage of target individuals who benefit from (or participate in) activities of each component (assessment of the acceptability of each component)
Intervention components' adaptation | Intervention components' implementation period
  Number of activities performed which have been modified to adapt them to the local context / total number of activities performed. A description of the adaptations performed will be provided. Data come from regular activity reports collected on a standardised form during components' implementation.
Satisfaction of target populations about the activities / tools, assessed by a 4-point Likert scale | End of the intervention components' implementation period
  Percentage of target individuals (adolescents, parents and general practitioners) who declare to be satisfied with each activity / tool (e.g., satisfaction of adolescents and school staff about the vaccination day organized inside the school premises, satisfaction of general practitioners about the e-learning training session). Satisfaction will be collected using self-administered (paper or online) questionnaires.

CONTACTS AND LOCATIONS:
Overall Officials: Nathalie THILLY, Pr, Principal Investigator — EA 4360 APEMAC - Université de Lorraine, Nancy; Serge GILBERG, Pr, Study Director — Département de Médecine Générale - Université Paris, Paris; Aurélie GAUCHET, Dr, Study Director — Université Grenoble Alpes, LIP/PC2S, EA 4145, Grenoble; Anne-Sophie LE DUC-BANASZUK, Dr, Study Director — Centre Régional de Coordination des Dépistages des cancers-Pays de la Loire, Angers; Amandine GAGNEUX-BRUNON, Dr, Study Director — GIMAP, EA 3064, Université Jean Monnet, Université de Lyon, Saint-Etienne, France; Karine CHEVREUL, Pr, Study Director — INSERM, ECEVE UMR 1123, Paris; Judith MUELLER, Dr, Study Director — Unité de Recherche et d'Expertise Epidémiologie des maladies émergentes, Institut Pasteur, Paris; Bruno GIRAUDEAU, Pr, Study Director — INSERM CIC 1415, CHRU de Tours, Tours, France
Locations (1):
- Secondary schools and GPs' practices of the participating municipalities, Multiple Locations, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Thilly N, Michel M, Simon M, Bocquier A, Gagneux-Brunon A, Gauchet A, Gilberg S, Le Duc-Banaszuk AS, Bruel S, Mueller JE, Giraudeau B, Chevreul K; PrevHPV Study Group. Effectiveness of a School- and Primary Care-Based HPV Vaccination Intervention: The PrevHPV Cluster Randomized Trial. JAMA Netw Open. 2024 May 1;7(5):e2411938. doi: 10.1001/jamanetworkopen.2024.11938. PMID 38780943
- [Result] Oudin Doglioni D, Gauchet A, Gagneux-Brunon A, Bruel S, Banaszuk AS, Thilly N, Sicsic J, Raude J, Mueller JE; PrevHPV Consortium. Shared human papillomavirus vaccine readiness within families: A psychometric analysis of parent-adolescent dyads in France. Health Psychol. 2024 Dec;43(12):893-903. doi: 10.1037/hea0001387. Epub 2024 Aug 22. PMID 39172389
- [Result] Bocquier A, Simon M, Michel M, Bonnay S, Adam I, Gilberg S, Bruel S, Gauchet A, LeDuc-Banaszuk AS, Gagneux-Brunon A, Mueller JE, Giraudeau B, Thilly N; PrevHPV Study Group. Implementation evaluation of a school- and primary care-based multicomponent intervention to improve HPV vaccine coverage: Results from the PrevHPV randomized controlled trial. J Infect Public Health. 2025 Nov;18(11):102931. doi: 10.1016/j.jiph.2025.102931. Epub 2025 Aug 15. PMID 40834467
- [Result] Dussault J, Gagneux-Brunon A, Le Duc-Banaszuk AS, Bruel S, Michel M, Gauchet A, Oudin Doglioni D, Sicsic J, Raude J, Barret AS, Thilly N, Mueller JE; PrevHPV Group. Effect of a multicomponent HPV intervention on self-reported HPV vaccine uptake and intention among French adolescents and parents: results from the national, cluster-randomised PrevHPV trial. BMJ Public Health. 2025 Aug 3;3(2):e001007. doi: 10.1136/bmjph-2024-001007. eCollection 2025. PMID 40761362
- [Result] Bocquier A, Michel M, Giraudeau B, Bonnay S, Gagneux-Brunon A, Gauchet A, Gilberg S, Le Duc-Banaszuk AS, Mueller JE, Chevreul K, Thilly N; PrevHPV Study group. Impact of a school-based and primary care-based multicomponent intervention on HPV vaccination coverage among French adolescents: a cluster randomised controlled trial protocol (the PrevHPV study). BMJ Open. 2022 Mar 24;12(3):e057943. doi: 10.1136/bmjopen-2021-057943. PMID 35332045
- [Derived] Bocquier A, Cadoret S, Fall E, Bonnay S, LeDuc-Banaszuk AS, Branchereau M, Gauchet A, Bruel S, Gagneux-Brunon A, Giraudeau B, Michel M, Mueller JE, Lefevre B, Thilly N; PrevHPV Study Group. Process evaluation of a school-based vaccination intervention to improve HPV vaccine coverage: A mixed-method study embedded in the French PrevHPV cluster randomized controlled trial. Vaccine. 2026 Feb 6;72:128122. doi: 10.1016/j.vaccine.2025.128122. Epub 2025 Dec 17. PMID 41412015